CLINICAL TRIAL: NCT07181785
Title: Single-center, Retrospective Study Aimed to Perform a Molecular Characterization of Aggressive B-cell Lymphomas (Diffuse Large B-cell Lymphoma, High-grade B-cell Lymphoma With MYC and BCL2 and/or BCL6 Translocations, High-grade B-cell Lymphoma Not Otherwise Specified) and to Observe the Clinical Patients' Outcomes According to the 2017 WHO Classification
Brief Title: Molecular Characterization and Outcomes of Aggressive B-Cell Lymphomas.
Acronym: CHARTHER
Status: Completed | Type: Observational
Sponsor: Andrés José Maria Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andrés José Maria Ferreri, MD & Prof., IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: CHARTHER
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult subjects (> 18 years old) of any age and gender affected by large B-cell lymphoma.: Histologically-confirmed diagnosis of LBCL (i.e., DLBCL, HGBCL, unclassifiable B-cell lymphoma with features intermediate between DLBCL and BL), or aggressive B-cell lymphomas with blastoid morphology (excluding blastoid variant of mantle cell lymphoma and lymphoblastic lymphoma)
  * Histopathological diagnosis performed between 2000 and 2019.
  * HIV sero-negativity
  * Age ≥18
  * Treatment with R-CHOP or other intensified polychemotherapy regimen
  * Availability of adequate histopathological samples at diagnosis for FISH analysis
  * Availability of clinical records and outcomes data
  Interventions: Combination Product: Treatments: anthracycline-based combinations followed or not by involved-field radiotherapy

INTERVENTIONS:
Combination Product: Treatments: anthracycline-based combinations followed or not by involved-field radiotherapy — Anthracycline-based combinations followed or not by involved-field radiotherapy

SUMMARY:
This is a retrospective analysis of the presence of chromosomal rearrangements involving MYC, BCL2 and BCL6 genes by FISH in a retrospective, single-center series of large B-cell lymphomas, in order to allow a better classifications of these cases according to the current WHO 2017 classification. If this evaluation will be confirmed as a reliable method to reclassify in different groups the evaluated tumors, it can be subsequently routinely apply to indicate the best treatment approaches in this high-risk setting of patients with a significant impact on patients' morbidity and mortality, and also on the health system and related costs.

ELIGIBILITY:
* Histologically-confirmed diagnosis of LBCL (i.e., DLBCL, HGBCL, unclassifiable B-cell lymphoma with features intermediate between DLBCL and BL), or aggressive B-cell lymphomas with blastoid morphology (excluding blastoid variant of mantle cell lymphoma and lymphoblastic lymphoma)
* Histopathological diagnosis performed between 2000 and 2019.
* HIV sero-negativity
* Age ≥18
* Treatment with R-CHOP or other intensified polychemotherapy regimen
* Availability of adequate histopathological samples at diagnosis for FISH analysis
* Availability of clinical records and outcomes data

Exclusion criteria

• Histologic diagnosis other than DLBCL or unclassifiable B-cell lymphoma with features intermediate between DLBCL and BL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (> 18 years old) of any age and gender affected by large B-cell lymphomas
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of pathologic diagnosis until death from any cause or last follow-up, whichever occurs first, assessed up to 60 months
  Overall survival (OS) is time from the date of pathologic diagnosis until death from any cause or last follow-up, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From the first day of treatment until relapse, progression, death , or last follow-up, whichever occurs first, assessed up to 60 months
  Progression-Free Survival (PFS) is the length of time during and after a disease treatment that a patient lives without the disease worsening or progressing
Overall Response Rate | From the first day of treatment until the date of first documented response assessment, typically within 6 months of treatment initiation
  the Overall Response Rate (ORR) measures the percentage of patients whose disease shows a reduction in size or is eliminated after a specific treatment. It includes patients who achieve either a Complete Response (CR), where all signs of the lymphoma disappear, or a Partial Response (PR), where there is a significant reduction in tumor burden but some signs of the disease remain
Duration of response (DOR; partial response [PR] + complete remission [CR]) | From the date of first documented response (CR or PR) until disease progression, relapse, death from any cause, or last follow-up, whichever occurs first, assessed up to 60 months
  Time from the date of first documented response (complete or partial) until disease progression, relapse, death from any cause, or last follow-up, whichever occurs first.
Relapse rates | From the date of first documented response (CR or PR) until disease relapse or last follow-up, whichever occurs first, assessed up to 60 months
  Proportion of patients who experience disease relapse after achieving a complete or partial response.
Relapse Pattern | From the date of first documented response (CR or PR) until disease relapse or last follow-up, whichever occurs first, assessed up to 60 months
  Description of the type and location of disease relapse, including nodal vs extranodal and local vs systemic recurrence
Incidence of chromosomal rearrangements involving MYC gene and BCL2 gene (so called "double hit lymphoma", representing 60% of HGBL) and/or BCL6 (also called "triple hit lymphoma", representing 20% of HG in Large B-cell Lymphomas. | At the time of pathologic diagnosis (baseline)
  Proportion of patients with documented genetic rearrangements of MYC, BCL2, or BCL6 detected at the time of pathologic diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT07181785/Prot_000.pdf